CLINICAL TRIAL: NCT06962657
Title: Mitigating Toxic Impact: The Role of Coenzyme Q10 in Post-Exposure Protection
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Beatrice Golomb, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 812491
Record Dates: First submitted 2025-04-05; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Toxicant Induced Chronic Multisymptom Illness and Associated Symptoms and Comorbidities
Keywords: Mixed toxic chemicals; Chronic multisymptom illness; Train derailment
MeSH Terms: interventions — Ubiquinone; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CoQ10 Arm (Active Comparator): Ubiquinone soft gel 100mg/3x day
  Interventions: Dietary Supplement: Ubiquinone 100 mg Oral Soft Gel
- Placebo Arm (Placebo Comparator): Soft gel placebo 3x/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ubiquinone 100 mg Oral Soft Gel — Active comparator arm receives three ubiquinone 100mg soft gels per day. Supplement is taken orally in divided doses, with the last soft gel not close to bedtime.
  Other Names: Coenzyme Q10
  Arms: CoQ10 Arm
Dietary Supplement: Placebo — Placebo comparator arm receives three placebo soft gels per day. Supplement is taken orally in divided doses, with the last soft gel not close to bedtime.
  Arms: Placebo Arm

SUMMARY:
This research study is being conducted to see if coenzyme Q10 (a nutritional supplement) might help to prevent and/or alleviate symptoms and health consequences and help to improve quality of life and physical function in residents affected by the February 2023 East Palestine, Ohio train derailment. This is a pilot study that is not powered to achieve benefit but seek to examine effect size and variance to aid in power calculations for a potential future better powered study.

ELIGIBILITY:
Inclusion Criteria:

* On Feb. 3, 2023, lived within 10 miles of the East Palestine, OH train derailment (closer in will receive preference). Others who were in the area for toxin mitigation and other reasons and show compatible symptoms will also be eligible.
* Meets Kansas symptom criteria for multi-symptom illness - originally defined for Gulf War Illness (has persistent symptoms, lasting greater than six months, that are of >mild severity in at least three of the six domains of fatigue/sleep, pain, neurological/cognitive/mood, gastrointestinal, respiratory and dermatologic). At least some symptoms must be new or worsened since the derailment.
* Access to internet and smart phone or computer for remote Qualtrics survey participation.
* Willing to perform the stipulated study elements.
* Took ≥80% of run-in soft gels.

Exclusion Criteria:

* Anticipated move from the area or other anticipated obstacle to participating for study duration.
* Participating in another clinical trial.
* Has a pre-existing health condition expected to produce significant and variable fluctuating symptoms (e.g. chronic infection and/or active cancer other than non-melanoma skin cancer).
* Contraindications to CoQ10, such as use of coumadin (although an interaction with CoQ10 is controversial).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
CoQ10 vs. placebo will (trend or effect) improve UCSD-20 (summed symptom score) | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  Number of symptoms (out of 20 on the UCSD Symptom Score Survey) showing more favorable change (trend or effect) on active treatment vs. on placebo. Outcomes are assessed as change from start of that treatment phase (from baseline for phase 1; and from 3 month crossover visit for phase 2).
CoQ10 vs. placebo will (trend or effect) improve GSRH | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  Mean change in single-item General Self-Rated Health (GSRH). Outcomes are assessed as change from start of that treatment phase (from baseline for phase 1; and from 3 month crossover visit for phase 2). 5 point scale, higher is good.
CoQ10 vs. placebo will (trend or effect) improve timed chair rises | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  Percent improved on timed chair rises from Gulf War Illness Modified Lower Extremity Summary Performance Score. Outcomes are assessed as change from start of that treatment phase (from baseline for phase 1; and from 3 month crossover visit for phase 2).

SECONDARY OUTCOMES:
Composite Adverse Health and Utilization Outcome 1 | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  CoQ10 vs. placebo will show (trend) improvement in dropouts for health related cause (e.g. not moved from area).
Composite Adverse Health and Utilization Outcome 2 | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  CoQ10 vs. placebo will show (trend) improvement in medical visits for cause (e.g. not routine annual follow up).
Composite Adverse Health and Utilization Outcome 3 | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  CoQ10 vs. placebo will show (trend) improvement in new health conditions/diagnoses/events.
Composite Adverse Health and Utilization Outcome 4 | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  CoQ10 vs. placebo will show (trend) improvement in new medications.
Relation of change in primary outcomes to change in blood level of coenzyme Q10 | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  We predict that greater rise in CoQ10 blood levels (in ug/mL) will be tied to greater improvement in primary endpoints.
Preferred treatment phase | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  More participants will "prefer" (perceive greater benefit from) the phase in which they received active (CoQ10) vs placebo treatment, assessed at still-blinded final visit (sign test).

OTHER OUTCOMES:
Mitochondrial function from blood spot card | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  Maximal respiration and spare capacity will be assessed by the "adopted transfer" technique. This uses Seahorse technology to look at mitochondrial function. Note this is an exploratory outcome, which means we will be exploring what can be seen, so it is not a primary or secondary aim.
Liver Function | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  Alanine aminotransferase and aspartate aminotransferase will be assessed as change from start of that treatment phase (from baseline for phase 1; and from 3 month crossover visit for phase 2) and compared on active treatment vs. placebo.
Inflammation (hsCRP) | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  Inflammation (hsCRP) will be assessed as change from start of that treatment phase (from baseline for phase 1; and from 3 month crossover visit for phase 2) and compared on active treatment vs. placebo.
Urine organic acids | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  Change in 8-OHdG will be more favorable (i.e. lower 8-OHdG) on active treatment than placebo. Urine organic acid abnormalities that relate to mitochondrial impairment (specifics of these will be different for different participants) will show favorable change on active treatment vs placebo.
AM salivary pH will be less acidic on CoQ10 than placebo | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
Salivary nitric oxide will be greater on active treatment than placebo | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
Urine pH will be less acidic on active treatment than placebo | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.
  Urine pH (preferred measurement time is at least 4 hours after the last meal -- ideally after lunch) will be less acidic on active treatment than placebo.
Change in peak flow will be more favorable on active treatment than placebo | Outcomes will be assessed at run-in (1-2 weeks before baseline) and baseline, and ~3 and ~6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice A. Golomb, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No